CLINICAL TRIAL: NCT04961879
Title: Comparative Study to Evaluate the Difference Between Reversed Cross Finger Flap Versus Reversed Island Homo-digital Flap in Distal Dorsal Finger Defect Reconstruction
Brief Title: Dorsal Finger Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elhossieny abdelaal mohamed, Principal Investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-07-09
Record Dates: First submitted 2021-07-13; First posted 2021-07-14 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Finger Injuries
MeSH Terms: conditions — Finger Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reversed Cross Finger Flap group 1 (Active Comparator)
  Interventions: Procedure: Reversed Cross Finger Flap
- Reversed island Homo-digital Flap group 2 (Active Comparator)
  Interventions: Procedure: reversed island homo-digital flap

INTERVENTIONS:
Procedure: Reversed Cross Finger Flap — distal dorsal finger defect will be reconstructed by reversed cross finger flap
  - reversed cross finger flap is a modified cross finger flap harvested from an adjacent finger .
  Arms: Reversed Cross Finger Flap group 1
Procedure: reversed island homo-digital flap — distal dorsal finger defect will be reconstructed by reversed island homo-digital flap
  - this flap is harvested from the same finger .
  Arms: Reversed island Homo-digital Flap group 2

SUMMARY:
objective of this study is To compare reversed cross finger flap with reversed island homo-digital flap in distal dorsal finger defect reconstruction regarding reliability & functional and aesthetic outcomes .

comparative study that will be conducted at Plastic surgery department, Sohag university hospital on 30 patients .The population of the study will be patients with distal dorsal digital defects. We will divide the cases into two equal groups: the first are operated with reversed cross-finger flap and the second are operated with reversed island homo-digital flap.

ELIGIBILITY:
Inclusion Criteria:

* patients with dorsal digital defect distal to distal interphalangeal joint (DIP) joint
* defect size ranged from 1 to 2 cm in width and 1-3 cm in length

Exclusion Criteria:

* chronic heavy smokers,
* traumatic injury to the donor site and perforator .

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
difference in range of motion between group 1 and group 2 | difference in range of motion between group 1 and group 2 will be measured at 4 months postoperative
  difference in range of motion between group 1 and group 2 will be measured by manual goniometer in degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt